CLINICAL TRIAL: NCT07212348
Title: The Effect of Laughter Yoga on Well-being and Psychological Adjustment in First-Year Midwifery Students: A Randomized Controlled Trial
Brief Title: Laughter Yoga in Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Rumeysa ÖZAYABAKAN, Asst. Prof., Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Agri Ibrahim Cecen University
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Well-Being, Psychological; Laughter Yoga
Keywords: Laughter Yoga; Well-being; Psychological Adjustment; Midwifery Students; adaption
MeSH Terms: conditions — Psychological Well-Being | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Students in the experimental group will participate in laughter yoga sessions conducted twice a week (Thursday and Friday) for four weeks, outside of class hours and in an indoor setting. The sessions will be carried out in subgroups of 9-10 students each, with a total of eight sessions. After completing the eight-session intervention, participants were sent reminder exercises via WhatsApp group for four weeks, and participants provided feedback with emojis as they practiced.
  Interventions: Behavioral: Laughter Yoga
- Control (No Intervention): Students in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Laughter Yoga — Students in the experimental group will participate in laughter yoga sessions conducted twice a week (Thursday and Friday) for four weeks, outside of class hours and in an indoor setting.
  Arms: Experimental

SUMMARY:
The aim of this study is to examine the effect of laughter yoga on well-being and psychological adjustment in first-year midwifery students and to evaluate its potential contributions in the context of adaptation to the educational process. The research is a randomized controlled experimental study. The study will be conducted at the Faculty of Health Sciences, Ağrı İbrahim Çeçen University.

The population of the study consists of all students newly enrolled in the Department of Midwifery, Faculty of Health Sciences, Ağrı İbrahim Çeçen University, in the 2025-2026 academic year. No sampling will be carried out; instead, all students who meet the inclusion criteria and volunteer to participate will be included in the study.

Participants will be randomly assigned to two groups: the experimental group (who will receive the laughter yoga intervention) and the control group (who will not receive any intervention). Thus, the study will be conducted as a randomized controlled experimental research.

The research data will be collected using the General Health Questionnaire, Student Information Form, Subjective Well-Being Scale, Psychological Well-Being Scale, and The Short Version of the Scales of General Well-Being.

DETAILED DESCRIPTION:
The study group consists of first-year students who started their studies in the Department of Midwifery, Faculty of Health Sciences, Ağrı İbrahim Çeçen University, in the fall semester of the 2025-2026 academic year. Participants will first be screened psychologically using the General Health Questionnaire-12 (GHQ-12). Students who are found not suitable for the study based on psychological screening will be excluded from the research.

Students included in the study will be randomly assigned to the experimental and control groups. Students in the experimental group will participate in laughter yoga sessions conducted twice a week (Thursday and Friday) for four weeks, outside of class hours and in an indoor setting. The sessions will be carried out in subgroups of 9-10 students each, with a total of eight sessions. Students in the control group will not receive any intervention.

Data will be collected at three points: pre-test (October 2025, before the intervention), post-test (November 2025, at the end of the fourth week of the intervention), and follow-up test (December 2025, one month after the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Newly enrolled in the Department of Midwifery, Faculty of Health Sciences, Ağrı İbrahim Çeçen University in the 2025-2026 academic year.
* Willing to participate in the study voluntarily.

Exclusion Criteria:

* İndividuals scoring 2 or higher on the GHQ-12.
* Those with urinary incontinence problems.
* Individuals who have recently undergone surgical operations.
* Those who regularly practice yoga, pilates, or similar sports/exercises.
* Individuals with asthma, COPD, or heart conditions.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire | At the time of study enrollment (baseline)
  The original version of the questionnaire, developed by David Goldberg in 1978, consists of 60 items and is used to determine the level of general psychopathology and to identify psychiatric cases in community surveys. All adaptations show high correlations with each other. .In this study, the GHQ-12, consisting of 12 items, was used. Each item asks about symptoms experienced over the past few weeks and has four response options: "not at all," "no more than usual," "rather more than usual," and "much more than usual." These four options are coded as 0 for "not at all," 1 for "no more than usual," 2 for "rather more than usual," and 3 for "much more than usual," or the administrator reads each item aloud and records the participant's response. In this study, the GHQ-type scoring used in Kılıç's (1996) validity and reliability study was applied. Therefore, participants with a GHQ-12 total score of 2 or higher are considered "cases requiring mental health assessment.
Student Information Form | At the time of study enrollment (baseline)
  Prepared by the researchers based on the literature, it includes questions such as age, parents' educational level, and voluntarily choosing the midwifery program.
Subjective Well-Being Scale | At baseline (pre-test), immediately after the intervention (post-test), and at 1-month follow-up
  Developed by Tuzgöl-Dost (2005), the scale aims to determine individuals' levels of subjective well-being by assessing their cognitive evaluations of life and the frequency and intensity of positive and negative emotions experienced. The scale consists of 46 items, 26 of which are positive and 20 negative statements. Negative items are reverse-scored. The total score ranges from 46 to 230, with higher scores indicating higher levels of subjective well-being. The scale uses a five-point Likert format: (5) Completely Agree, (4) Mostly Agree, (3) Partially Agree, (2) Slightly Agree, and (1) Strongly Disagree. To assess reliability, Cronbach's alpha coefficient and the test-retest method were used. Cronbach's alpha reliability coefficient was found to be 0.93, and the test-retest reliability for the entire scale was 0.86. For validity, confirmatory factor analysis showed factor loadings between 0.32 and 0.63.
Psychological Well-Being Scale | At baseline (pre-test), immediately after the intervention (post-test), and at 1-month follow-up
  The Psychological Well-Being Scale was developed by Diener and colleagues (2009-2010) to complement existing well-being measures and to assess socio-psychological well-being. The Turkish adaptation of the scale was conducted by Telef (2011; 2013).
  Items on the Psychological Well-Being Scale are rated on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). All items are positively worded. Total scores range from 8 (if a respondent answers "strongly disagree" to all items) to 56 (if a respondent answers "strongly agree" to all items). Higher scores indicate that the individual possesses multiple psychological resources and strengths.
The Short Version of the Scales of General Well-Being | At baseline (pre-test), immediately after the intervention (post-test), and at 1-month follow-up
  The Short Version of the Scales of General Well-Being (SVSGW) was developed by Longo, Coyne, and Joseph. The validity and reliability of the Turkish version of this scale were established by Kalafatoğlu and Balcı Çelik. The scale is a single-factor instrument consisting of 13 items rated on a five-point Likert scale. The minimum possible score on the scale is 13 and the maximum score is 65. Higher scores indicate a higher level of general well-being. The Cronbach's alpha coefficient of the original scale was reported as 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Rumeysa ÖZAYABAKAN, Asst. Prof., Study Director — Agri Ibrahim Cecen University; Betül UNCU, Principal Investigator — İstanbul University-Cerrahpaşa; Ebru SOLMAZ, Principal Investigator — Agri Ibrahim Cecen University
Locations (1):
- Ağrı İbrahim Çeçen Üniversitesi, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes